CLINICAL TRIAL: NCT05909189
Title: LEADing Dementia End-of-Life Planning Conversations
Acronym: LEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kara Dassel, Professor, Assistant Dean, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GRANT13319762; 5R01AG069033-03 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-06-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: advance care planning; caregiving; decision-making
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The LEAD Intervention is a web-baed platform that integrates the LEAD Guide with self-paced educational modules that guide care recipient-care partner pairs through conversations and the process of dementia-focused advance care planning. The aims of this study are: 1. To describe the acceptability, usability, and feasibility of the LEAD Intervention. Methods: Conduct a process evaluation using survey-based outcome assessments and qualitative analysis of participant-recorded advance care planning conversation(s)to identify facilitators and/or barriers to intervention participation. 2. To assess the initial efficacy of the LEAD Intervention on the primary outcome and secondary outcomes as perceived by both the care recipient and the care partner. 3. To examine advance care planning congruence as a mechanism of action for the LEAD Intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADRD dyads (Experimental): This is a single-arm study enrolling 60 ADRD community-based dyads.
  Interventions: Other: LEADing Dementia End-of-Life Planning Conversations

INTERVENTIONS:
Other: LEADing Dementia End-of-Life Planning Conversations — The LEAD Intervention is self-administered and delivered through an interactive, web-based platform designed according to recommended functionalities and user-designed principles. Through three distinct modules, the LEAD Intervention will facilitate the advance care planning processes of 1) defining care recipients' values and preferences for care, 2) developing advance care planning congruence within the pair, or a shared understanding of the care recipient's values and preferences, through conversation(s), and 3) encouraging ongoing advance care planning conversation and documentation that can be shared beyond the pair. All modules will include video tutorials to introduce the goals and tasks as well as provide interactive resources to provide support and education relevant to the content of each module. The three modules are intended to be followed in a sequential pattern.

SUMMARY:
Advance care planning is important for all adults, but perhaps even more so for the 5.7 million persons with Alzheimer's disease or related dementia (ADRD), due to the progressive and protracted cognitive deterioration associated with the disease process. In the context of ADRD, medical decision-making at the end of life is typically left to one's care partner, who often does not have the knowledge or confidence in their ability to make such decisions. This study will refine and evaluate a web-based platform, called the LEAD Intervention (Life-Planning in Early Alzheimer's and other Dementias), which is designed to help persons in the preclinical or early stage of ADRD engage in conversations about, document, and share their end-of-life values and preferences with a care partner, extended family members, and health care providers.

DETAILED DESCRIPTION:
Advance care planning is the process that allows individuals to express their future healthcare values and preferences so that these wishes can be enacted in the event that they become incapacitated and unable to participate in their own healthcare decisions. In the case of Alzheimer's disease or related dementia (ADRD), the person with dementia (care recipient), almost inevitably loses decisional capacity toward the end of life, given the progressive decline in cognitive functioning that accompanies the disease over time. The care partners to persons with dementia, most often family members such as spouse/partners and adult children, are therefore tasked with making end-of-life decisions on behalf of the care recipient with ADRD. These care partners are not always well-informed of the care recipient's end-of-life values and preferences and therefore may not feel confident in their ability to make decisions regarding care and treatment at the end-of-life, resulting in unnecessary, futile, and often unwanted medical treatments and interventions. Oftentimes, families do not want to engage in these challenging conversations and wait too long, whereby the care recipient with ADRD no longer has the decisional ability to participate in the advance care planning process. We developed "The LEAD Guide" (Life-Planning in Early Alzheimer's and other Dementias), as a tool to help persons with preclinical awareness of ADRD risk and those with early-stage cognitive impairment to begin these important conversations with a care partner. In this NIH Stage-1 behavioral intervention study we will refine the LEAD Intervention based on our pilot work (Stage 1A) and then evaluate the usability, acceptability, feasibility, and initial efficacy of the LEAD Intervention (Stage 1B). We will recruit a diverse sample of 60 community-dwelling ADRD pairs, defined as a care recipient in the preclinical or early stage of ADRD, plus their current or anticipated care partner (i.e., spouse/partner or adult child). Results are expected to show that the LEAD Intervention can improve outcomes related to decision-making self-efficacy through greater advance care planning congruence and improve subjective well-being, anxiety, and relationship quality as perceived and reported by both the care recipient and the care partner. Results from this study have the potential to guide and accelerate the implementation of the LEAD Intervention in community and healthcare practice, where a dementia-focused advance care process is needed.

ELIGIBILITY:
Inclusion Criteria:

* Care Recipient (CR) is age 50+
* CR Is interested in having conversations about and documenting wishes for future end-of-life care
* CR has noticed changes in memory or thinking skills indicative of preclinical or early stage of AD, OR
* CR has been diagnosed with mild cognitive impairment, Alzheimer's disease, or another type of dementia and in the preclinical or early stage
* Care Partner (CP) is age 18+
* CP is a Spouse/partner, family member, or close friend of CR

Exclusion Criteria:

* Has moderate to severe symptoms of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Decision-Making Self-Efficacy | Week 20
  Decision-making efficacy as measured by both the care recipient and care partner as measured by the Family Decision-Making Self-Efficacy Scale

SECONDARY OUTCOMES:
Relationship Quality | Week 20
  Relationship quality as measured by both the care recipient and care partner as measured by the Dyadic Relationship Scale (DRS)
Anxiety | Week 20
  Perceived symptoms of anxiety by both the care recipient and care partner as measured by the PROMIS Emotional Distress-Anxiety-Short Form 8a
Subjective well-being | Week 20
  Perceived subjective well being of care recipient and care partner as measured by the PROMIS General Life Satisfaction- Short Form 5a

CONTACTS AND LOCATIONS:
Overall Officials: Kara Dassel, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We welcome analysis and use by other investigators once our primary aims have been analyzed and disseminated. All data and resources will be shared following the policies of the University of Utah and NIH. We will share LEAD intervention survey data by depositing these data at National Alzheimer's Coordinating Center (NACC), which is an NIH-funded repository. These data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes such as examining components of self-efficacy. Data will be shared in an Excel file format that will allow for easy access to qualified users. Shared data will include participant demographic information and survey data relevant to all predictor and primary study outcome variables.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon completion of the study and once findings have been published by the study team.
Access Criteria: We will share LEAD intervention survey data by depositing these data at National Alzheimer's Coordinating Center (NACC), which is an NIH-funded repository.

REFERENCES:
- [Background] Dassel KB, Utz R, Supiano K, McGee N, Latimer S. The Influence of Hypothetical Death Scenarios on Multidimensional End-of-Life Care Preferences. Am J Hosp Palliat Care. 2018 Jan;35(1):52-59. doi: 10.1177/1049909116680990. Epub 2016 Dec 17. PMID 28273753
- [Background] Supiano KP, McGee N, Dassel KB, Utz R. A Comparison of the Influence of Anticipated Death Trajectory and Personal Values on End-of-Life Care Preferences: A Qualitative Analysis. Clin Gerontol. 2019 May-Jun;42(3):247-258. doi: 10.1080/07317115.2017.1365796. Epub 2017 Oct 9. PMID 28990872
- [Background] Dassel K, Utz R, Supiano K, Bybee S, Iacob E. Development of a Dementia-Focused End-of-Life Planning Tool: The LEAD Guide (Life-Planning in Early Alzheimer's and Dementia). Innov Aging. 2019 Aug 2;3(3):igz024. doi: 10.1093/geroni/igz024. eCollection 2019 Jul. PMID 31392286
- [Derived] Clayton JL, Utz RL, Aruscavage N, Bybee SG, Bigger SE, Iacob E, Dassel KB. Using community engagement with FRAME: Framework for reporting adaptations and modifications to evidence-based interventions. Contemp Clin Trials Commun. 2024 Nov 26;42:101398. doi: 10.1016/j.conctc.2024.101398. eCollection 2024 Dec. PMID 39717518